CLINICAL TRIAL: NCT05922605
Title: Analgesic Effects of Caudal S-ketamine for Supplementation of Ropivacaine Caudal Analgesia in Children With Hypospadias
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Associate Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Caudal S-ketamine
Record Dates: First submitted 2023-06-15; First posted 2023-06-28 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Analgesia; S-ketamine; Pediatrics; Caudal Block; Hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Esketamine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Patients allocated to study groups using computer generates random list & group assignment is sealed in sequentially numbered opaque envelopes that open after induction of anesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Experimental): the children are given a mixture of 0.2%ropivacaine 0.7 ml／kg and preservative-free S-ketamine 0.5 mg/kg for caudal analgesia.
  Interventions: Drug: S-ketamine & Ropivacaine
- Group C (Active Comparator): The children are given 0.2%ropivacaine 0.7 ml／kg and saline of equal volume caudally.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: S-ketamine & Ropivacaine — The experiment group (Group E) will receive a mixture of ropivacaine 0.2% 0.7 ml／kg and preservative-free S-ketamine 0.5 mg/kg caudally for postoperative analgesia.
  Arms: Group E
Drug: Ropivacaine — The experiment group (Group C) will receive ropivacaine 0.2% 0.7 ml／kg plain and equial volume saline caudally for postoperative analgesia.
  Arms: Group C

SUMMARY:
Caudal analgesia with ropivacaine is commonly used in sub-umbilical pediatric surgery. However, increasing the dosage of ropivacaine has not been found to prolong the action significantly while complications will be serious.

Ketamine as an additive to caudal administration had been shown to prolong the duration of postoperative analgesia, while the analgesic effectiveness of S-ketamine, the S(+)-enantiomer of ketamine with less possibility to induce psychomotor disturbances, is not clear. In this prospective randomized double-blind clinical trial , the investigators aimed to study the effect of S-ketamine as additive on the duration of caudal analgesia.

DETAILED DESCRIPTION:
Forty-four children scheduled for hypospadias randomize into 2 groups. Group E (n=22) (0.2% ropivacaine 0.7 ml／kg and S-ketamine 0.5 mg/kg), group C(n=22)( 0.2%ropivacaine 0.7ml／kg and equivalent saline) intraoperative and postoperative hemodynamics will be recorded. Postoperative pain is assessed using an established 6-item FLACC score at 1h,3h,6h,12h,24h,48h, or the time when children complain of pain after surgery. A score of more15μg/kg is administered.Investigators propose to compare the duration of caudal analgesia provided by plain ropivacaine and by a mixture of ropivacaine and S-ketamine.

ELIGIBILITY:
Inclusion Criteria:

* informed parent consent, ASA I or II children, between 3months and 18 years of age,and weighing <28kg, scheduled for elective hypospadias surgery with general anesthesia will be recruited.

Exclusion Criteria:

* Patients who have congenital abnormalities of lower spine and meninges.
* Patients with hypersensitivity to any local anesthetics
* Children with coagulation disorders
* Presence of Infections at puncture sites
* Preexisting neurological disease
* Refusal to consent by parent/guardian

Ages: 3 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
duration of caudal analgesia | 48 hours after the caudal injection
  Duration of analgesia is defined as the time from caudal injection to the first need for systemic analgesia.

SECONDARY OUTCOMES:
morphine consumption | 48 hours after caudal block
  The Face, Legs, Activity, Cry, and Consolability (FLACC) scale at 1 hour (h), 3h,6h,12h,24h,48h or the time when children complain of pain after surgery. A score of more than 3 points is taken as an indication of inadequate analgesia and morphine 15ug/kg was administered .
FLACC score | 48 hours after the caudal block
  The Face, Legs, Activity, Cry, and Consolability (FLACC) scale
complication | 48 hours after the caudal block
  the incidence of residual motor block, urinary retention, paraesthesia; the incidence of respiratory depression ,vomiting ,nystagmus ,pruritus，odd behavior;.the sedation scores etc.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, M.D., Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunes Y, Secen M, Ozcengiz D, Gunduz M, Balcioglu O, Isik G. Comparison of caudal ropivacaine, ropivacaine plus ketamine and ropivacaine plus tramadol administration for postoperative analgesia in children. Paediatr Anaesth. 2004 Jul;14(7):557-63. doi: 10.1111/j.1460-9592.2004.01220.x. PMID 15200652
- [Background] De Negri P, Ivani G, Visconti C, De Vivo P. How to prolong postoperative analgesia after caudal anaesthesia with ropivacaine in children: S-ketamine versus clonidine. Paediatr Anaesth. 2001 Nov;11(6):679-83. doi: 10.1046/j.1460-9592.2001.00742.x. PMID 11696143
- [Background] Weber F, Wulf H. Caudal bupivacaine and s(+)-ketamine for postoperative analgesia in children. Paediatr Anaesth. 2003 Mar;13(3):244-8. doi: 10.1046/j.1460-9592.2003.01018.x. PMID 12641687
- [Background] Martindale SJ, Dix P, Stoddart PA. Double-blind randomized controlled trial of caudal versus intravenous S(+)-ketamine for supplementation of caudal analgesia in children. Br J Anaesth. 2004 Mar;92(3):344-7. doi: 10.1093/bja/aeh076. Epub 2004 Jan 22. PMID 14742331
- [Background] Koinig H, Marhofer P, Krenn CG, Klimscha W, Wildling E, Erlacher W, Nikolic A, Turnheim K, Semsroth M. Analgesic effects of caudal and intramuscular S(+)-ketamine in children. Anesthesiology. 2000 Oct;93(4):976-80. doi: 10.1097/00000542-200010000-00017. PMID 11020749
- [Background] Brenner L, Marhofer P, Kettner SC, Willschke H, Machata AM, Al-Zoraigi U, Lundblad M, Lonnqvist PA. Ultrasound assessment of cranial spread during caudal blockade in children: the effect of different volumes of local anaesthetics. Br J Anaesth. 2011 Aug;107(2):229-35. doi: 10.1093/bja/aer128. Epub 2011 Jun 3. PMID 21642642
- [Background] Narasimhan P, Kashyap L, Mohan VK, Arora MK, Shende D, Srinivas M, Kashyap S, Nath S, Khanna P. Comparison of caudal epidural block with paravertebral block for renal surgeries in pediatric patients: A prospective randomised, blinded clinical trial. J Clin Anesth. 2019 Feb;52:105-110. doi: 10.1016/j.jclinane.2018.09.007. Epub 2018 Sep 19. PMID 30243061